CLINICAL TRIAL: NCT03927547
Title: Sleep Disordered Breathing and Cardiopulmonary Disease in Peruvian Highlanders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00170895; R34HL135360 (NIH)
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-03

CONDITIONS: Sleep Disordered Breathing; Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Subjects will undergo sleep study in subjects' randomized sleep posture. Randomization will be recorded separately from sleep study recordings. These recordings will be reviewed by trained sleep study technicians who will be blinded to randomization. Blood samples will also be assayed for markers of glucose control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inclined Sleep (Experimental): Inclined mattress at 15 degrees
  Interventions: Device: Inclined Sleep
- Flat Sleep (No Intervention): Plane mattress

INTERVENTIONS:
Device: Inclined Sleep — Study participants randomized to the interventional arm will be instructed to sleep on inclined wedge mattress.
  Other Names: wedge mattress; postural therapy
  Arms: Inclined Sleep

SUMMARY:
Overall objective: To understand the feasibility of performing a randomized trial using a simple, minimally-invasive postural therapy approach to improve sleep disordered breathing (SDB).

DETAILED DESCRIPTION:
Specific Aims:

* To examine the relative efficacy of postural therapy (a 15-degree wedge mattress) on measures of chronic cardiometabolic stress in high altitude residents.
* To determine the tolerability of postural therapy.

Primary outcomes, at 4 and 8 weeks:

* Mean nocturnal oxyhemoglobin saturation (SPO2)
* Apnea-hypopnea index (AHI).

Secondary outcomes

* Markers of hypoxemia exposure: the investigators will evaluate for differences in average hemoglobin and erythropoietin concentrations between intervention groups using t-tests or Wilcoxon rank sum tests, as considered appropriate. If transformations are necessary, the investigators will use Box-Cox power transform to identify the best transformation for the investigators' data.
* Markers of metabolic dysfunction: the investigators will evaluate for differences in average Glycated hemoglobin test (HbA1c), homeostatic model assessment of insulin resistance (HOMA-IR), total cholesterol, low-density lipoprotein cholesterol (LDL), High-density lipoprotein cholesterol (HDL), triglycerides, SVEGF-R1 , and soluble Vascular Endothelial Growth Factor (SVEGF-1) concentrations between intervention groups using t-tests or Wilcoxon rank sum tests, as appropriate. If transformations are necessary, the investigators will use Box-Cox power transform to identify the best transformation for the investigators' data.
* Markers of cardiometabolic stress: the investigators will evaluate for differences in average systolic blood pressure (SBP), diastolic blood pressure (DBP), pulse, and % change in endothelial function (reactive hyperemia index) as assessed by brachial artery reactivity testing (BART) between intervention groups using t-tests or Wilcoxon rank sum tests, as considered appropriate.
* Adherence (the average number of nights during the 8-week period that participants slept on the wedge mattress),

ELIGIBILITY:
Inclusion criteria

* Age 40-80 years
* Daytime oxyhemoglobin saturation ≥80%, seated.
* Body mass index ≥25 kg/m2
* Hemoglobin >13 g/dL in women and >15 g/dL in men
* Ability to provide informed consent
* Sleeps at home in same bed every night
* Expected stable residence for at least 6 months
* Sleeps with two pillows or fewer
* Demonstrate acute improvement in SDB severity with postural therapy
* Able to sleep ≥5 hours at an incline for all three nights during the run-in period

Exclusion criteria

* Works the night-shift or a rotating shift
* Has an indication or preference for sleeping upright, semi-recumbent or at an incline
* Chronic insomnia or a non-respiratory sleep disorder
* Physician-established diagnosis of diabetes, lung, cardiovascular, liver, or chronic kidney disease
* Using home oxygen therapy or other respiratory assistive device [e.g., continuous positive airway pressure (CPAP), nebulizer]
* Self-reported severe gastrointestinal reflux
* Self-report of occult blood or history of gastrointestinal bleeding in the past 3 months
* Pregnancy
* Unable to sleep ≥5 hours at an incline for all three nights during the run-in period

The following exclusion criteria apply only for those undergoing spirometry for safety reasons. Participants with any one of these criteria, will be excluded from spirometry but can still participate in the rest of the screening phase:

* Surgery of the heart, chest, lungs in the past 3 months (participants will be revisited at a later period)
* Heart attack in the past 3 months (participants will be revisited at a later period)
* History of eye surgery
* History of abdominal surgery in the past 3 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-09-29 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Respiratory Disturbance Index (RDI) | Baseline, 4 weeks, 8 weeks
  The investigators will measure a change in Respiratory Disturbance Index (RDI) defined as an oxygen desaturation of at least 4 percent associated with autonomic signs of arousal. Specifically, autonomic arousals are defined as concurrent rises in heart rate and attenuation of arterial tonometry.
  Normal < 5 percent 5 percent < Mild < 15 percent 15 percent < Moderate < 30 percent Severe > 30 percent
Change in Mean oxyhemoglobin saturation (percent) during sleep | Baseline, 4 weeks, 8 weeks
  The investigators will measure mean oxyhemoglobin saturation (%SaO2) during sleep as assessed by WatchPAT home sleep study at baseline and week 8.

SECONDARY OUTCOMES:
Tolerability of postural therapy as assessed by adherence monitor | 2, 4, 6 and 8 weeks
  Adherence monitor will measure sleep over the set time points and tolerability is defined as a recorded time on the wedge for a minimum of 5 hours.
Change in average plasma hemoglobin concentration (g/dL) | Baseline, 8 weeks
Change in average Glycated hemoglobin test (HbA1c) | Baseline, 8 weeks
  This will measure percentage (%) of HbA1c in the blood.
Change in serum erythropoietin (EPO) concentration | Baseline, 8 weeks
  The concentration of EPO in the sample is expressed in International Units per litre (U/L) and is determined by calibration against a reference standard.
Change in soluble Vascular Endothelial Growth Factor (SVEGF-1) concentrations | Baseline, 8 weeks
  Plasma levels of SVEGF-1 (pg/mL)
Change in homeostatic model assessment of insulin resistance (HOMA-IR) | Baseline, 8 weeks
  Units of measurement is mass units.
Change in total plasma cholesterol level (mg/dL) | Baseline, 8 weeks
Change in plasma low-density lipoprotein (LDL) cholesterol level (mg/dL) | Baseline, 8 weeks
Change in plasma high-density lipoprotein (HDL) cholesterol level (mg/dL) | Baseline, 8 weeks
Change in plasma triglyceride concentration (mg/dL) | Baseline, 8 weeks
Change in Vascular endothelial growth factor receptor 1 (SVEGF-R1) concentration | Baseline, 8 weeks
  Units of measurement pg/mL
Change in mean blood pressure (mmHg) | Baseline, 8 weeks
Change in Brachial Artery Reactivity Testing (BART) assessment | Baseline, 8 weeks
  Assessed by endothelial function using high-frequency ultrasound visualized brachial artery reactivity testing. Endothelial function is characterized by flow-mediated vasodilation of the brachial artery, which is measured by comparing the brachial artery diameter at rest to the diameter after increased forearm blood flow (reactive hyperemia).
  Unit of measurement is mass units.

CONTACTS AND LOCATIONS:
Overall Officials: William Checkley, Principal Investigator — Johns Hopkins University
Locations (1):
- Prisma Org, Puno, Peru

IPD SHARING:
Plan to Share IPD: Undecided